CLINICAL TRIAL: NCT05858632
Title: Immune Spatial Features of Guselkumab Cutaneous Response
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-35862
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis of Scalp
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guselkumab treatment (Experimental): Guselkumab treatment for ~ 9 months
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab treatment for ~ 9 months

SUMMARY:
This study examines the effect of IL-23 blockade with Guselkumab on the immune cells of scalp psoriasis lesions.

DETAILED DESCRIPTION:
This is a one-arm, open-label study to examine the effect of Guselkumab . Guselkumab is a FDA-approved medication for the treatment of psoriasis. This study will examine how Guselkumab affects immune cells within scalp psoriasis lesions. Ten subjects with moderate to severe scalp psoriasis will be enrolled. Biopsy samples will be collected and undergo molecular profiling to correlate profiles with Guselkumab treatment response.

ELIGIBILITY:
Inclusion Criteria: possess a PSSI (psoriasis scalp severity index) of ≥12

Exclusion Criteria:

1. taking systemic immunosuppressives in the last 4 weeks
2. pregnancy
3. severe immunodeficiency (either from genetic or infectious causes).
4. tuberculosis or other active serious infection
5. active systemic malignancy.
6. breast-feeding
7. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
8. Males who are trying to conceive

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in psoriasis scalp severity index score (PSSI) | baseline and 9 months
  PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. PSSI scores will be taken pre- and mid-treatment. Scores range from 0 to 72, with higher scores indicating more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No